CLINICAL TRIAL: NCT05740657
Title: Evaluation of Opioids and Metabolites in Hair and Sweat of Pediatric Patients in a Monitored Clinical Context, by Means of Targeted Liquid Chromatography-tandem Mass Spectrometry
Brief Title: Observational Study on the Incorporation of Opioids and Their Metabolites Into Hair of Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01693
Record Dates: First submitted 2023-01-31; First posted 2023-02-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use, Unspecified
Keywords: hair analysis; fentanyl; fentalogs; new synthetic opioids; opioids
MeSH Terms: interventions — Fentanyl; Remifentanil; Sufentanil; Hydromorphone; Oxycodone; Morphine; Alfentanil; Nalbuphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples Without DNA — Hair samples (without hair root) Sweat Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- KISPI 000: Patients of the group received one or multiple clinically approved opioids, namely; Fentanyl, Remifentanil, Sufentanil, Alfentanil, Oxycodone, Morphine, Nalbuphine, Hydromorphone and Methadon. The drugs were administered in the course of a surgery or for pain management.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — The drugs were administered in the course of a surgery or for pain management.
  Other Names: Remifentanil; Sufentanil; Hydromorphone; Oxycodone; Morphine; Alfentanil; Nalbuphine; Methadon

SUMMARY:
Hair analysis is a well-established and important tool in both forensic and clinical context. When it comes to the interpretation of positive hair analysis results, reliable and comprehensive reference data is essential. Such data on opioids, especially novel synthetic ones (such as fentanyl and its analogues (fentalogs)) is currently highly limited. This applies especially to hair with pediatric origin, due to differences in the metabolism and hair anatomy in children compared to adults.

Investigators hypothesize that opioids, both traditional and novel synthetic ones exhibit detectable concentrations and distinct metabolite ratios within the hair matrices of pediatric patients. Thus, this observational, prospective research study provides 150 hair and sweat samples from children who received opioids as part of surgery or pain management. The samples will be consecutively extracted and analyzed using a sensitive targeted liquid chromatography-tandem mass spectrometry (LC-MS/MS) method, enabling the quantitative determination of the opioid and metabolite concentrations. The study thereby contributes valuable reference data for both forensic and clinical applications, addressing challenges in interpreting hair analysis results in especially pediatric populations. Further, a deeper understanding of the mechanisms (e.g. via sweat) and pharmacokinetic processes involved in the opioid incorporation to hair will be achieved. The study has received ethical approval from the Swiss Ethics Board (approval number: 2022-01693 / amendment approval date: 09.01.2024).

ELIGIBILITY:
Inclusion Criteria:

* Obtained written informed-consent from legal representatives (and oral consent from the patient).
* Patient's age must be within date of birth irrespective of gestational age to completed 13th year of life
* Patients that received single or multiple treatment (either with single doses or continuous infusion) of fentanyl, remifentanil or sufentanil either during surgery or during stay in the pediatric intensive care unit

Exclusion Criteria:

* Patient's age of 14 or older
* Inability to understand the study procedure due to language or cognitive reasons (applies to legal representatives and elder children)
* Denied or missing informed consent
* Insufficient amount of head hair to obtain hair sample
* Cosmetic hair treatment, like coloring, bleaching and dying

Ages: 1 Day to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of patients (newborns, infants, children and adolescents up to 13 years of age) from the pediatric intensive care unit from the Children's Hospital Zurich. Patients in focus are exposed to fentanyl and fentalogs (remifentanil, sufentanil and alfentanil) or other more traditional opioids (such as morphine, oxycodone and methadone) either during surgery or as part of post-operative pain management for up to three months prior to study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the opioid and metabolite concentrations (pg/mg: units of picograms of opioid per milligram hair) in the hair samples of the study population. | Through study completion, an average of two years
  For the collected hair samples, a two-stage extraction is performed, using methanol and a buffered methanol-water mixture for 90 minutes each. The extracts are then evaporated, resuspended in a 3:7 mixture of methanol and eluent A (20 mM ammonium formate with 0.1% (v/v) formic acid in water). The hair sample extracts will then be measured on an the LC-MS/MS system (SCIEX Triple Quad™ 7500 LC-MS/MS (QTRAP) System).
  A validated analysis method will be used for the analysis of the following opiates, opioids or their metabolites: hydromorphone, 4-ANPP, acetylcodeine, acetylmorphine, alfenanil, betahydroxyfentanyl, codeine, dihydrocodeine, fentanyl, hydrocodone, methadone, morphine, naloxone, norfentanyl, norsufentanil, omegahydroxyfentanyl, oxycodone, oxymorphone, pethidine, remifentanil, remifentanil-acid, sufentanil and tramadol. The data is processed with the software SciexOS version 1.6.7.
Evaluation of the opioid and metabolite concentrations (ng/mL: units of nanograms of opioid per milliliter) in the sweat extracts of the study population. | Through study completion, an average of two years
  The extraction procedure of the sweat swabs looks as follows: the cotton ends of the forensic swabs will be cut and extracted with methanol. The methanol extracts will then be diluted to avoid detector saturation and mixed in a 3:7 ratio with eluent A. The sweat sample extracts will then be measured on an the LC-MS/MS system (SCIEX Triple Quad™ 7500 LC-MS/MS (QTRAP) System).
  A validated analysis method will be used for the analysis of the following opiates, opioids or their metabolites: hydromorphone, 4-ANPP, acetylcodeine, acetylmorphine, alfenanil, betahydroxyfentanyl, codeine, dihydrocodeine, fentanyl, hydrocodone, methadone, morphine, naloxone, norfentanyl, norsufentanil, omegahydroxyfentanyl, oxycodone, oxymorphone, pethidine, remifentanil, remifentanil-acid, sufentanil and tramadol. The data is processed with the software SciexOS version 1.6.7.

SECONDARY OUTCOMES:
Normative opioid concetration values and metabolite reatios in pediatric hair. | after data evaluation, 3 months after end of study
  This data will be analyzed by using descriptive statistics (box plots) including the median, mean, 10th percentile, and 90th percentile values and for their distribution (normal or non-normal) by Shapiro-Wilks Test. Thus, opioid specific concentration values and metabolite ratios in hair of children will be established.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Binz, Principal Investigator — University Zürich; Florian Zapf, Dr., Principal Investigator — University's Children Hospital
Locations (1):
- University's Children Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The outcomes of the research will be published in peer-reviewed journals. Data will be strictly anonymized.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: starting after publication
Access Criteria: upon request via e-mail